CLINICAL TRIAL: NCT03209518
Title: Special Drug Use Surveillance of Leuplin PRO for Injection Kit 22.5 mg in "Premenopausal Breast Cancer"
Brief Title: Special Drug Use Surveillance of Leuprorelin for Injection Kit 22.5 mg in "Premenopausal Breast Cancer"
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: Leuprorelin-5003; JapicCTI-163203 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2017-07-04; First posted 2017-07-06 (Actual); Results first posted 2019-11-01 (Actual); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Premenopausal Breast Cancer
MeSH Terms: interventions — Leuprolide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Leuprorelin acetate: Usually, for adults, 22.5 mg of Leuprorelin acetate was subcutaneously administered once every 24 weeks. Refer to the Precautions section of the package insert. Participants received Leuprorelin as part of routine medical care.
  Interventions: Drug: Leuprorelin acetate

INTERVENTIONS:
Drug: Leuprorelin acetate — Leuplin PRO for Injection Kit 22.5 mg
  Other Names: Leuplin PRO for Injection Kit 22.5 mg

SUMMARY:
The purpose of this survey is to evaluate the safety in patients with premenopausal breast cancer receiving Leuprorelin in the routine clinical setting.

DETAILED DESCRIPTION:
The drug being tested in this survey is called Leuprorelin for Injection Kit 22.5 mg. Leuprorelin is being tested to treat people who have premenopausal breast cancer.

This survey will look at the safety in patients with premenopausal breast cancer receiving the drug in the routine clinical setting.

The survey will enroll approximately 300 patients.

- Leuprorelin

This multi-center survey will be conducted in Japan.

ELIGIBILITY:
Inclusion Criteria:

- Participants with premenopausal breast cancer will be included.

Exclusion Criteria:

* Participants with a history of hypersensitivity to any ingredients of Leuplin PRO, synthesized LH-RH, or LH-RH analogues
* Pregnant or potentially pregnant participants and breastfeeding participants

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The survey population will consist of participants with a diagnosis of premenopausal breast cancer and received dose of Leuprorelin for Injection Kit 22.5 mg in the routine medical care.
Sampling Method: Non-Probability Sample
Enrollment: 312 (Actual)
Dates: Start 2016-03-18 (Actual); Primary Completion 2018-10-10 (Actual); Study Completion 2018-10-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Takeda selected site, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No
Takeda makes patient-level, de-identified data sets and associated documents available for all interventional studies after applicable marketing approvals and commercial availability have been received (or program is completely terminated), an opportunity for the primary publication of the research and final report development has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the survey at 52 investigative sites in Japan, from 18 March 2016 to 10 October 2018.
Pre-assignment Details: Participants with a historical diagnosis of premenopausal breast cancer were enrolled. Participants received Leuprorelin as part of routine medical care.
Groups:
- Leuprorelin Acetate 22.5 mg: Usually, for adults, 22.5 mg of Leuprorelin acetate was subcutaneously administered once every 24 weeks. Refer to the Precautions section of the package insert. Participants received Leuprorelin as part of routine medical care.
Period: Overall Study
Arm/Group | Leuprorelin Acetate 22.5 mg
Started | 312
Completed | 310
Not Completed | 2
Not completed — Case Report Forms Uncollected | 1
Not completed — Protocol Deviation | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set, The safety analysis set was defined as participants who were evaluable for the safety without major protocol deviation within those who administered the survey drug.
Arm/Group | Leuprorelin Acetate 22.5 mg
Number analyzed (Participants) | 310
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.8 (5.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 310
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: Participants]
  Japan | 310
Duration between Diagnosis of Premenopausal Breast Cancer and Survey Start [Mean (Standard Deviation); unit: Months] — Mean duration between the first diagnosis of premenopausal breast cancer and the start of the survey was reported.
  Months | 23.80 (20.777)
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — Number of participants with each score of ECOG Performance Status at the survey start was reported. Following are ECOG grades. 0:Fully active, perform all pre-disease activities without restriction. 1:Restricted in physically strenuous activity but ambulatory, carry out work of a light or sedentary nature. 2:Ambulatory, capable of self-care, unable to carry out any work activities, up and about more than (>) 50% of waking hours. 3:Capable of limited self-care, confined to bed or chair >50% of waking hours. 4:Completely disabled, not capable of any self-care, totally confined to bed or chair.
  Participants
    0 | 302
    1 | 8
Target of Treatment [Count of Participants; unit: Participants]
  Participants with Neoadjuvant Therapy | 14
  Participants with Adjuvant Therapy | 272
  Participants with Progressive Breast Cancer | 12
  Participants with Recurrent Breast Cancer | 12
Number of Participants with Hormone Receptor Expression [Count of Participants; unit: Participants] | 310
Healthcare Category [Count of Participants; unit: Participants] — Participants were categorized as outpatient and inpatient.
  Participants
    Outpatient | 308
    Inpatient | 2
Predisposition to Hypersensitivity [Count of Participants; unit: Participants] — Number of participants who had or did not have a liability or tendency to suffer from hypersensitivity was reported.
  Participants
    Had No Predisposition to Hypersensitivity | 282
    Had Predisposition to Hypersensitivity | 26
    Unknown | 2
Medical Complications [Count of Participants; unit: Participants] — Complications defined as a disease or a health condition for each participant at the start of study. Complications were classified as congenital anomalies, endocrine disorders, hematologic disorders, psychiatric and nervous system disorders, cardiovascular disorders, respiratory disorders, gastrointestinal (GI) disorders, renal disease and other complications. Other complications included all complications except for those mentioned above.
  Participants
    Had No Medical Complications | 267
    Had Medical Complications | 43
Medical History of Thromboembolism [Count of Participants; unit: Participants] — Number of participants with or without medical history of thromboembolism was reported.
  Participants
    Had No Medical History of Thromboembolism | 307
    Had Medical History of Thromboembolism | 3
Height [Mean (Standard Deviation); unit: Centimeters (cm)] — Population: The number analyzed is the number of participants with data available for analysis.
  Centimeters (cm)
    number analyzed (Participants) | 290
    (all) | 159.4 (5.26)
Weight [Mean (Standard Deviation); unit: Kilograms (kg)] — Population: The number analyzed is the number of participants with data available for analysis.
  Kilograms (kg)
    number analyzed (Participants) | 290
    (all) | 55.55 (10.650)
BMI [Mean (Standard Deviation); unit: kg/meter(m)^2] — Body Mass Index = weight (kg)/[height (m)^2] Population: The number analyzed is the number of participants with data available for analysis.
  kg/meter(m)^2
    number analyzed (Participants) | 289
    (all) | 21.86 (3.952)
Prior Treatment with LH-RH Agonists [Count of Participants; unit: Participants] — Number of participants who were treated or were not treated with LH-RH agonists for premenopausal breast cancer was reported.
  Participants
    Not Treated with Drugs | 77
    Treated with LH-RH Agonists | 233
Prior Treatment with Drugs for Premenopausal Breast Cancer [Count of Participants; unit: Participants] — Number of participants who were treated or were not treated with drugs except LH-RH agonists for premenopausal breast cancer was reported.
  Participants
    Not Treated with Drugs | 47
    Treated with Drugs | 263

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Had One or More Adverse Events
Time Frame: Up to Week 24
Population: as for baseline characteristics
Measure: Number; unit: Percentage of Participants
Arm/Group | Leuprorelin Acetate 22.5 mg
Number analyzed (Participants) | 310
Percentage of Participants | 6.45

2. Secondary Outcome: Percentage of Participants Who Had One or More Adverse Reactions
Description: Adverse drug reaction refers to adverse events related to the administered drug.
Time Frame: Up to Week 24
Population: as for baseline characteristics
Measure: Number; unit: Percentage of Participants
Arm/Group | Leuprorelin Acetate 22.5 mg
Number analyzed (Participants) | 310
Percentage of Participants | 5.48

ADVERSE EVENTS:
Time Frame: Up to Week 24
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to survey treatment.
Arm/Group | Leuprorelin Acetate 22.5 mg
All-Cause Mortality (participants affected / at risk) | 0/310
Serious Adverse Events (participants affected / at risk) | 0/310
Other Adverse Events (participants affected / at risk) | 20/310
OTHER ADVERSE EVENTS (reported when occurring in more than 0.5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Leuprorelin Acetate 22.5 mg (N=310)
Hot flush (Vascular disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Injection site induration (General disorders) | 4
Injection site pain (General disorders) | 9
Injection site pruritus (General disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2019-04-05): https://cdn.clinicaltrials.gov/large-docs/18/NCT03209518/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-04): https://cdn.clinicaltrials.gov/large-docs/18/NCT03209518/SAP_001.pdf